CLINICAL TRIAL: NCT07342621
Title: SMASH: Study to Evaluate the Clinical Efficacy of an Extensively Hydrolysed Infant Formula With Synbiotics and a Human Milk Oligosaccharide (HMO) in Infants With Cow's Milk Protein Allergy (CMPA)
Acronym: SMASH
Status: Recruiting | Type: Observational
Sponsor: Outcomes'10 (Network)
Responsible Party: Sponsor
Other Study IDs: NUT-2023-185-APLV
Record Dates: First submitted 2025-11-20; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cow's Milk Protein Allergy (CMPA); Food Hypersensitivity; Infant Nutrition Disorders; Gut Microbiota
Keywords: Extensively Hydrolyzed Formula; Synbiotics; Cow's Milk Protein Allergy; Real World Evidence; Microbiota; Gastrointestinal Symptoms
MeSH Terms: conditions — Milk Hypersensitivity; Food Hypersensitivity; Infant Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants with suspected or confirmed CMPA

SUMMARY:
Cow's milk protein allergy (CMPA) is one of the most common food allergies in infants, with an estimated prevalence between 2% and 5%. The number of diagnosed cases has increased in recent years, with clinical manifestations involving the gastrointestinal tract, respiratory system, skin, or systemic reactions. Dietary elimination of cow's milk protein remains the mainstay of treatment, using extensively hydrolyzed formulas (EHF) or amino acid-based formulas (AAF), depending on the severity of the allergy.

This study aims to evaluate the clinical effect, as reported by physicians, of an extensively hydrolyzed whey-based formula (Almirón Pepti Syneo®) containing a symbiotic mixture (scGOS/lcFOS 9:1 and Bifidobacterium breve M-16V), the human milk oligosaccharide 2'-fucosyllactose (2'-FL), and a reduced amount of purified lactose, in infants with suspected or confirmed CMPA in a real-world clinical practice setting.

This is a prospective, longitudinal, open-label, single-arm, multicenter study including approximately 41 infants under 10 months of age at several primary care centers and one hospital in Valencia, Spain. Each participant will be followed for four weeks. A subgroup of participants will also provide stool samples to explore the effect of the study formula on gut microbiota composition.

DETAILED DESCRIPTION:
Background and Rationale

Cow's milk protein allergy (CMPA) is a frequent condition in pediatric populations and a major cause of medical consultation during early infancy. Although prevalence estimates vary across studies, it is generally reported between 2% and 5%. CMPA can present with cutaneous, gastrointestinal, respiratory, or systemic symptoms and may impact growth, nutritional status, and family quality of life.

The cornerstone of management is dietary elimination of cow's milk protein. In infants requiring formula feeding, extensively hydrolyzed formulas (EHF) or amino acid-based formulas (AAF) are recommended, depending on allergy severity. Recent evidence suggests that gut microbiota composition plays a key role in the development and modulation of allergic diseases, and that prebiotics, probiotics, and synbiotics may beneficially modulate immune responses via the gut microbiome.

Almirón Pepti Syneo® is an extensively hydrolyzed whey-based formula that includes a symbiotic mixture (scGOS/lcFOS 9:1 and Bifidobacterium breve M-16V), the human milk oligosaccharide 2'-fucosyllactose (2'-FL), and a reduced content of purified lactose. Previous studies have demonstrated its safety, efficacy in managing CMPA symptoms, and support for adequate infant growth.

Objectives

Primary Objective:

- To evaluate the effect of an extensively hydrolyzed formula containing synbiotics and 2'-FL on physician-reported outcomes related to CMPA symptoms (cutaneous, respiratory, gastrointestinal, and/or systemic) in infants with suspected or confirmed CMPA.

Secondary Objectives:

* To assess parent- or caregiver-reported outcomes related to CMPA symptoms.
* To evaluate the impact of the infant's condition on parental or caregiver quality of life.
* To describe infant growth during the study period.
* To assess parental acceptability and satisfaction with the study product.

Exploratory Objective:

- To explore the effect of the study formula on gut microbiota composition and stool characteristics in infants with suspected or confirmed CMPA.

Study Design

This is a prospective, longitudinal, open-label, single-arm, multicenter study conducted at approximately 13 primary care centers and one hospital (Hospital Quirón, Valencia, Spain). The study will enroll 41 infants under 10 months of age with suspected or recently confirmed CMPA.

Each infant will be followed for four weeks after the initiation of the study formula. Parents or legal guardians will complete standardized and ad hoc questionnaires regarding symptom evolution, gastrointestinal function, and product acceptability, while investigators will record clinical and anthropometric data using an electronic case report form (eCRF).

A subgroup of infants whose parents or guardians consent to the exploratory stool analysis will provide samples for microbiota assessment, processed at the sponsor's laboratories in Singapore and Utrecht.

Sample Size and Study Population

A total of 41 infants under 10 months of age with suspected or recently diagnosed CMPA will be recruited, assuming a 30% potential dropout rate. Infants with prior use of EHF, AAF, rice hydrolysate, or soy formulas will be excluded.

Variables

Collected data will include:

* Sociodemographic and baseline characteristics: sex, birth weight and length, gestational age, family history of allergy, feeding type, and antibiotic use.
* Anthropometric measures: weight, length, and head circumference at baseline and study end.
* Clinical assessments: CoMiSS, SCORAD, and IGSQ-13 scores.
* Parent-reported outcomes: ad hoc symptom and stool questionnaires, PO-SCORAD, FAQL-PB, and acceptability/satisfaction surveys.
* Safety: adverse events and concomitant medications.

Study Duration

Recruitment will take place over approximately nine months. Each participant will be followed for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Infants under 10 months of age at study start (Visit 1).
* Suspected or recently confirmed cow's milk protein allergy (CMPA), as determined by the investigator.
* Already formula-fed, or parents/legal guardians have decided to initiate formula feeding.
* Inclusion in the study coincides with the first prescription of a hypoallergenic formula.
* Written informed consent obtained from parents or legal guardians in accordance with local regulations.

Exclusion Criteria:

* Infants with functional gastrointestinal symptoms in whom atopy or food allergy is not suspected.
* Infants who have previously used an extensively hydrolyzed formula (EHF), an amino acid-based formula (AAF), a rice hydrolysate formula, or a soy-based formula.
* Infants who have previously used a partially hydrolyzed formula for the prevention of cow's milk protein allergy (CMPA).
* Infants for whom an amino acid-based formula (AAF) is more appropriate as first-line management, including severe forms of CMPA.
* Contraindications to the use of synbiotics (e.g., preterm infants <40 weeks of corrected gestational age at study start, immunodeficiency, short bowel syndrome, parenteral nutrition, post-pyloric feeding, central venous catheter, oncology treatment, or graft-versus-host disease).
* Any other condition, as assessed by the investigator, that contraindicates the use of an extensively hydrolyzed formula.
* Any other circumstance, as assessed by the investigator, indicating that the parents or legal guardians are not capable of complying with the study procedures.

Max Age: 10 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants under 10 months of age with suspected or recently confirmed cow's milk protein allergy (CMPA) who are initiating the use of a hypoallergenic formula as part of routine clinical management. All participants will receive an extensively hydrolyzed whey-based formula containing synbiotics and 2'-fucosyllactose (2'-FL) and will be followed prospectively for four weeks.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in investigator-reported allergy symptom scores | Baseline (Visit 1) and Week 4 (Visit 2)
  Change from baseline to Week 4 in investigator-assessed allergy symptoms in infants with suspected or confirmed cow's milk protein allergy, measured using four validated or ad hoc instruments:

SECONDARY OUTCOMES:
Change in parent-reported allergy symptom scores from baseline to Week 4 | Baseline and Week 4
  Change in parent- or caregiver-reported symptoms Differences between baseline and Week 4 will be analyzed and categorized according to improvement (reduction in score) or no improvement.
Change in stool characteristics from baseline to Week 4 | Baseline and Week 4
  Parent-reported stool characteristics (consistency and color). Frequencies of stool types will be summarized for each visit, and changes over time will be described.
Change in parental quality of life related to infant allergy from baseline to Week 4 | Baseline and Week 4
  Change in the Food Allergy Quality of Life-Parental Burden Questionnaire (FAQL-PB) score from baseline to Week 4. Improvement will be defined as a reduction in the total score. Descriptive statistics and frequencies of improvement will be presented.
Change in infant anthropometric z-scores from baseline to Week 4 | Baseline and Week 4
  Change in z-scores for weight, length, and head circumference calculated according to World Health Organization (WHO) growth standards. Differences between baseline and Week 4 will be summarized using descriptive statistics.
Parental acceptability and satisfaction with the study formula | At Week 4
  Parent- or caregiver-reported acceptability and satisfaction with the study product. Frequencies of responses and consumption ratios (prepared vs. consumed product) will be summarized, and temporal trends will be described.

OTHER OUTCOMES:
Changes in gut microbiota composition after 4 weeks of formula use | Baseline and Week 4
  Stool microbiota composition assessed through 16S rRNA gene sequencing (and optional metagenomics in a subset). Outcomes include relative abundance of Bifidobacterium spp. and Bifidobacterium breve, microbiota composition (beta diversity, stability, or maturation index), microbial diversity (alpha diversity), and differential abundance of bacterial taxa from phylum to species levels.
Changes in microbial metabolites in stool samples | Baseline and Week 4
  Concentrations and relative proportions of short-chain fatty acids levels in stool samples, measured by laboratory analysis.
Changes in microbial metabolites in stool samples | Baseline and Week 4
  Concentrations and relative proportions of ammonia levels in stool samples, measured by laboratory analysis.
Changes in stool pH | Baseline and Week 4
  Stool pH measured at baseline and Week 4 as an indicator of gut microbial activity and metabolic profile.

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (12):
  - Quironsalud Valencia Hospital, Valencia, Valencia
  - Trinitat Health centre, Valencia, Valencia
  - Malva-rosa Health centre, Valencia, Valencia
  - República Argentina Health centre, Valencia, Valencia
  - Salvador Pau Health centre, Valencia, Valencia
  - Serrería 2 Health Centre, Valencia, Valencia
  - Serrería I Health Centre, Valencia, Valencia
  - Trafalgar Health centre, Valencia, Valencia
  - Miguel Servet Health centre, Valencia, Valencia
  - Alboraya Health centre, Valencia, Valencia
  - Cañada Health centre, Valencia, Valencia
  - Eliana Health centre, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No